CLINICAL TRIAL: NCT05786131
Title: Complete Revascularization Versus Culprit Lesion Only PCI in NSTEMI (-COMPLETE-NSTEMI-)
Brief Title: Complete Revascularization Versus Culprit Lesion Only PCI in NSTEMI
Acronym: CompleteNSTEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leipzig Heart Science gGmbH (Other)
Collaborators: Heart Center Leipzig at University of Leipzig (Unknown); German Federal Ministry of Education and Research (Other Government); IHF GmbH - Institut für Herzinfarktforschung (Other); Stiftung IHF - Institut für Herzinfarktforschung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-019
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Non-ST-elevation Myocardial Infarction; Multivessel Coronary Artery Disease
Keywords: NSTEMI; Multivessel coronary artery disease; culprit-lesion only PCI; multivessel percutaneous coronary intervention
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- culprit-lesion-only revascularization (Experimental): Patients will receive optimal medical therapy without further revascularization of non-culprit lesions (neither during index hospitalization nor during follow-up). Angina pectoris will be treated medically as recommended in the chronic coronary syndrome guidelines. Revascularization of non-culprit lesions will only be permitted if at least one bailout criteria is met.
  Interventions: Procedure: Culprit-lesion revascularization
- multivessel complete revascularization (Experimental): Patients will receive complete revascularization of all angiographically significant non-culprit lesions, either during the index procedure, the index hospitalization, or staged within 45 days after PCI of the culprit lesion.
  Interventions: Procedure: Culprit-lesion revascularization; Procedure: Non-culprit-lesion revascularization

INTERVENTIONS:
Procedure: Culprit-lesion revascularization — Percutaneous coronary intervention of culprit-lesion
  Other Names: Culprit-lesion PCI
Procedure: Non-culprit-lesion revascularization — Complete percutaneous coronary intervention of all angiographically significant non-culprit lesions
  Other Names: multivessel PCI
  Arms: multivessel complete revascularization

SUMMARY:
Prospective, randomized, controlled, multicenter, open-label trial to study whether multivessel percutaneous coronary intervention (PCI) is superior over culprit-lesion only PCI in patients with non-ST-segment elevation myocardial infarction (NSTEMI) and multivessel coronary artery disease.

DETAILED DESCRIPTION:
The complete revascularization versus culprit lesion only PCI in NSTEMI (COMPLETE-NSTEMI) trial aims to investigate whether multivessel complete PCI is superior over culprit-lesion only PCI in patients with NSTEMI and multivessel coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* NSTEMI as suggested by high-sensitivity troponin algorithms
* Multivessel coronary artery disease
* Identifiable culprit lesion
* Informed consent

Exclusion Criteria:

* Age <18 years
* Cardiogenic shock
* Sustained ventricular tachycardia (VT) or ventricular fibrillation (VF)
* Contraindication for coronary revascularization
* Prior coronary artery bypass graft
* Indication for coronary artery bypass graft surgery
* Non-culprit lesion located in the left main coronary artery
* Co-morbidity with life expectancy less than 6 months
* Type 2 myocardial infarction
* Pregnancy and breast feeding period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3390 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Composite rate of cardiovascular death or rehospitalization for non-fatal myocardial infarction | During follow-up (2 years estimated average duration)

SECONDARY OUTCOMES:
Rate of Cardiovascular death | During follow-up (2 years estimated average duration)
Rate of Rehospitalization for non-fatal myocardial infarction | During follow-up (2 years estimated average duration)
Rate of all-cause death | During follow-up (2 years estimated average duration)
Rate of ischemia-driven revascularization | During follow-up (2 years estimated average duration)
Rate of rehospitalization for heart failure | During follow-up (2 years estimated average duration)
Composite rate of all-cause death, rehospitalization for non-fatal myocardial infarction, or rehospitalization for ischemia-driven revascularization | During follow-up (2 years estimated average duration)
Rate of coronary artery bypass surgery | During follow-up (2 years estimated average duration)
Quality of Life (EQ-5D-5L) | 12 months
  European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) Score 1-5 for each dimension, 1 means best outcome EQ VAS score between 0 and 100; higher score means better outcome
Rate of bleeding | 6 months
Rate of stroke | 6 months
  Ischemic and Hemorrhagic
Rate of contrast-induced acute kidney injury | 6 months
  AKIN grade I-III
Rate of coronary procedure-related myocardial infarction | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, MD, Prof. Dr., Study Chair — Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology
Locations (58):
- Austria (3):
  - LKH Univ. Klinikum Graz, Clinical Department of Cardiology, Graz
  - Medizinische Universität Innsbruck, Universitätsklinik für Innere Medizin III, Innsbruck
  - Klinik Ottakring, 3. medizinische Abteilung, Vienna
- Germany (55):
  - Zentralklinik Bad Berka, Klinik für Kardiologie, Bad Berka
  - Universitäts-Herzzentrum Bad Krozingen, Klinik für Kardiologie und Angiologie, Bad Krozingen
  - Kerckhoff Klinik, Bad Nauheim
  - Herz- und Diabeteszentrum NRW, Universitätsklinikum der Ruhr-Universität Bochum, Klinik für Allgemeine und Interventionelle Kardiologie/Angiologie, Bad Oeynhausen
  - BG Klinikum Unfallkrankenhaus Berlin gGmbH, Klinik für Innere Medizin/Kardiologie, Berlin
  - Charité - University Medicine Berlin, Department of Internal Medicine and Cardiology, Campus Virchow Klinikum, Berlin
  - Klinikum Bielefeld gem. GmbH, Klinik für Kardiologie und Internistische Intensivmedizin, Bielefeld
  - Klinik für Kardiologie und Rhythmologie, St. Josef Hospital, Universitätsklinikmum der Ruhr-Universität Bochum, Bochum
  - Klinikum Links der Weser, Innere Medizin II, Bremen
  - Städtisches Klinikum Dessau; Klinik für Innere Medizin II (Kardiologie, Angiologie, Diabetologie, internistische Intensivmedizin), Dessau
  - St. Johannes Hospital, Klinik für Innere Medizin I, Dortmund
  - Herzzentrum Dresden GmbH, Universitätsklinik an der Technischen Universität Dresden, Klinik für Innere Medizin und Kardiologie, Dresden
  - Heinrich Heine Universitätsklinikum Düsseldorf Institut für Kardiologie, Pneumologie und Angiologie, Düsseldorf
  - HELIOS Klinikum Erfurt, Medizinische Klinik III - Kardiologie, Erfurt
  - Universitätsklinikum Erlangen, Medizinische Klinik 2, Erlangen
  - Elisabeth Krankenhaus Essen, Klinik für Kardiologie und Angiologie, Essen
  - Universitätsklinikum Essen, Klinik für Kardiologie und Angiologie, Essen
  - Universitätsklinikum Freiburg, Klinik für Kardiologie und Angiologie, Freiburg im Breisgau
  - Klinikum Fulda, Medizinischen Klinik 1 - Kardiologie, Angiologie und Intensivmedizin, Fulda
  - Universitätsklinikum Gießen und Marburg GmbH, Medizinische Klinik I, Kardiologie, Giessen
  - University Medical Center Göttingen, Department of Cardiology and Pneumology, Georg-August University, Göttingen
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Innere Medizin B, Greifswald
  - Universitätsklinikum Halle (Saale), Klinik für Innere Medizin III, Halle
  - Asklepios Klinik St. Georg, Kardiologie und Internistische Intensivmedizin, Hamburg
  - Universitäres Herz- und Gefäßzentrum UKE Hamburg GmbH, Klinik für Kardiologie, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Klinik für Kardiologie, Angiologie und Pneumologie, Medizinische Klinik 3, Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Klinik für Innere Medizin II, Homburg
  - Universitätsklinikum Jena, Klinik für Innere Medizin I, Kardiologie, Angiologie, Internistische Intensivmedizin, Jena
  - Vincentius-Diakonissen-Kliniken gAG Medizinische Klinik III, Kardiologie, Intensivmedizin, Angiologie, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Klinik für Innere Medizin III mit den Schwerpunkten Kardiologie und internistische Intensivmedizin, Kiel
  - Asklepios Klinik Langen, Abteilung Medizinische Klinik I, Langen
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Kardiologie, Leipzig
  - Klinikum St. Georg gGmbH Klinik für Kardiologie und Internistische Intensivmedizin, Leipzig
  - Heart Center Leipzig at University of Leipzig, Department of Internal Medicine/Cardiology, Leipzig
  - Klinikum der Stadt Ludwigshafen, Medizinische B Klinik, Ludwigshafen
  - Universitätsklinikum Schleswig Holstein, Medizinische Klinik II, Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg, Klinik für Kardiologie und Angiologie, Magdeburg
  - Brüderklinikum Julia Lanz, Theresienkrankenhaus, Mannheim
  - Universitätsmedizin Mannheim, I. Medizinische Klinik, Kardiologie, Angiologie, Hämostaseologie und Internistische Intensivmedizin, Mannheim
  - Universitätsklinikum Gießen und Marburg GmbH - Standort Marburg, Klinik für Innere Medizin - Kardiologie, Angiologie und Intensivmedizin, Marburg
  - Klinikum der Universität München, Medizinische Klinik und Poliklinik I, München
  - Deutsches Herzzentrum München, Klinik für Herz- und Kreislauferkrankungen, München
  - Klinikum Neumarkt, Neumarkt
  - Klinikum Nürnberg, Medizinische Klinik 8 - Schwerpunkt Kardiologie, Universitätsklinik der Paracelsus Medizinischen Privatuniversität, Nuremberg
  - Universitätsklinik für Kardiologie am Klinikum Oldenburg, Oldenburg
  - Helios Vogtland-Klinikum Plauen, Plauen
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Innere Medizin II, Regensburg
  - Universitätsmedizin Rostock, Zentrum für Innere Medizin, Abteilung für Kardiologie, Rostock
  - Helios Kliniken Schwerin, Klinik für Kardiologie und Angiologie, Schwerin
  - Krankenhaus der Barmherzigen Brüder Trier, Herzzentrum Innere Medizin III - Kardiologie, Trier
  - Universitätsklinikum Tübingen, Medizinische Klinik, Innere Medizin III, Kardiologie und Angiologie, Tübingen
  - Schwarzwald-Baar Klinikum VS, Studienteam Kardiologie, Villingen-Schwenningen
  - Städtisches Klinikum Wolfenbüttel gGmbH, Klinik für Innere Medizin - Kardiologie,, Wolfenbüttel
  - Helios Klinikum Wuppertal, Herzkreislaufforschung, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feistritzer HJ, Jobs A, Zeymer U, Schneider S, Lauten P, Ferenc M, Weferling M, Brinkmann R, Winkler S, Landmesser U, Trippel T, Stellbrink C, Wienbergen H, Furnau G, Mollmann H, Linke A, Jung C, Lauten A, Achenbach S, Rassaf T, Schmitz T, Cremer S, Olivier C, Schachinger V, Sossalla S, Toischer K, Templin C, Sedding D, Clemmensen P, Tigges E, Meincke F, Sharar HA, Kulenthiran S, Schulze PC, Jacobshagen C, Frank D, Baldus S, Lehmann R, Spies C, Klein N, Eitel I, Zahn R, Schmeisser A, Gori T, Lurz P, Akin I, Chatzis G, Rizas K, Kessler T, Ademaj F, Elsasser A, Maier L, Oner A, Staudt A, Werner N, Geisler T, Kessler M, Ferrari MW, Seyfarth M, Nordbeck P, Ewen S, Bietau C, Haghikia A, Reinstadler SJ, Geppert A, Hosler N, Toth-Gayor G, Billmann B, Tschierschke R, Schmidt C, Fichtlscherer S, Thiele H; COMPLETE-NSTEMI Investigators. Complete revascularization versus culprit-lesion only PCI in patients with NSTEMI and multivessel disease - Design and rationale of the randomized COMPLETE-NSTEMI trial. Am Heart J. 2025 Sep;287:94-106. doi: 10.1016/j.ahj.2025.04.007. Epub 2025 Apr 8. PMID 40209841